CLINICAL TRIAL: NCT04034914
Title: A Preliminary Pilot Study to Tailor and Evaluate the Feasibility of Child and Parent Yoga (CAPY) During Chemotherapy Infusion
Brief Title: Yoga Intervention in Supporting Children With Cancer and Their Parents During Chemotherapy Infusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Sheila Ridner, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC SUPP 1935; NCI-2019-04525 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2019-07-17; First posted 2019-07-26 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Therapy (Experimental)
  Interventions: Other: Questionnaire administration

INTERVENTIONS:
Other: Questionnaire administration — Ancillary studies

SUMMARY:
This trial studies how well Yoga works in supporting children with cancer and their parents during chemotherapy infusion. Pediatric cancer and its treatment is one of life's most stressful events for children and their parents. Yoga is an ancient holistic healing science that incorporates postures, breathing, relaxation, and meditation to facilitate harmony between body, mind, and spirit. Participating in Yoga exercise may improve the negative psychosocial effects in children with cancer and their parents during chemotherapy treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To determine the feasibility of Yoga for children with cancer and their parents, specifically
* Identify possible required modifications for safe and feasible practice during infusions.
* Obtain recruitment estimates and determine barriers.
* Assess satisfaction.

SECONDARY OBJECTIVES:

* To determine the feasibility of administering and acceptability of measures to assess preliminary efficacy of Yoga for the following outcomes:
* Child psychological distress (stress, anxiety).
* Parent psychological distress (stress, anxiety, anger, depression).
* Child and parent physiological stress (heart rate, respiratory rate, and blood pressure).
* Parent-child communication.
* Child physical symptoms.

OUTLINE:

Patients and parents participate in up to 8 Yoga sessions consisting of check in, awareness, breathing practices, gentle movement, and relaxation over 30 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Children: 8-17 years of age, within 4 weeks of: 1) any new cancer diagnosis or newly diagnosed relapsed cancer, and 2) medical clearance who anticipate 3-weeks of continous contact with Monroe Carell Jr. Children's Hospital.
* Parents: 18 years of age and older, child's primary caregiver (planning to attend appointments, infusions visits, or be in hospital rooms/clinics) or secondary caregiver (an as needed back-up to primary).

Children and Parents: able to speak and understand English, absence of cognitive impairment, and willing to engage in Yoga as part of a dyad.

Exclusion Criteria:

* CHILDREN: Medical conditions that would prohibit the safe implementation of a Yoga practice
* PARENTS: Practices Yoga weekly
* PARENTS: Pregnant or plans to become pregnant during next 3 months
* CHILDREN AND PARENTS: Unwilling to work as a dyad.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Modifications | Up to 2 years
  Will be assessed qualitatively. A tally of the specific modifications will be maintained to determine if particular modification are made more frequently than others.
Recruitment | Up to 2 years
  The total number of eligible child-parent dyads approached to achieve an enrolled sample of 5 dyads will be tallied.
Retention | Up to 2 years
  The number of the enrolled child-parent dyads who complete both the self-report assessments required at baseline (T1 - prior to first Yoga session), the Yoga protocol, and the measures at the end-of-infusion (T2 - prior to last Yoga session) will be tallied. The proportion completing will be used to inform the level of over-recruitment required in future studies of efficacy.
Barriers | Up to 2 years
  Participants who do not complete the study will be contacted and queried as to the reason for the lack of completion. A tally of the specific barriers will be maintained to determine if particular barriers are encountered more frequently than others. This information will inform possible modifications required to the protocol in future research.
Participant satisfaction | Up to 2 years
  The total number of responses to the 14 satisfaction questions with a rating > 4 (maximum rating = 7) will be generated for each of the 5 parent participants. It is expected that all participants will exceed that threshold for all questions. If not, frequency distributions will be used to summarize the responses to each of the 14 items to assess which produced the lower ratings. Responses to open-ended questions will be analyzed qualitatively. Findings from both components of the satisfaction survey (program satisfaction and yoga survey) will be used to revise the Yoga protocol as needed.

SECONDARY OUTCOMES:
Child psychological distress | Up to 2 years
  Will assess child distress using Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Psychological Stress Experiences- Short Form
Parent psychological distress | Up to 2 years
  Will assess parent distress using the PROMIS Depression - Short Form
Parent psychological distress | Up to 2 years
  Will assess parent distress using the PROMIS Emotional Distress - Anger - Short Form
Parent psychological distress | Up to 2 years
  Will assess parent distress using the PROMIS Anxiety
Child and parent physiological stress | Up to 2 years
  Will assess blood pressure
Child and parent physiological stress | Up to 2 years
  Will assess heart rate
Child and parent physiological stress | Up to 2 years
  Will assess respiratory rate
Parent-child communication | Up to 2 years
  Will be assessed using the Parent-Adolescent Communication Scale (PACS). Participants answer 20-40 questions. A total score is calculated ranging from 20-100 with higher scores indicating more positive communication.
Child physical symptoms | Up to 2 years
  Will be assessed using the PROMIS Pediatric Physical Stress Experiences -Short Form.
Parent psychological distress | Up to 2 years
  Parent distress will be assessed using the NIH Toolbox Perceived Stress
Child psychological distress | Up to 2 years
  Child distress will be assessed using the PROMIS Pediatric Anxiety - Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Ridner, PhD, Principal Investigator — Vanderbilt University School of Nursing; Terrah Akard, PhD, Principal Investigator — Vanderbilt University School of Nursing
Locations (1):
- Vanderbilt University School of Nursing, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No